CLINICAL TRIAL: NCT06689566
Title: Evaluating Metabolic and Anti-inflammatory Effect of Genistein on Post-myocardial Infarction Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202404082RIND
Record Dates: First submitted 2024-11-04; First posted 2024-11-14 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Myocardial Infarction (MI)
Keywords: inflammation
MeSH Terms: conditions — Myocardial Infarction; Inflammation | interventions — Genistein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- genistein group (Experimental)
  Interventions: Dietary Supplement: genistein

INTERVENTIONS:
Dietary Supplement: genistein — the patients will receive genistein 250mg BID orally for complete 3 months. Afterwards, there will be 3 months washout period. Patients would then be followed for outcome measurement.

SUMMARY:
The goal of this clinical trial is to learn if genistein works to provide a beneficial effect to show lipid lowering effect and anti-inflammatory effects and slow the progression of atherosclerosis in post-myocardial infarction adults. It will also learn about the safety of genistein. The main questions it aims to answer are:

Does genistein lower triglyceride in participants? What medical problems do participants have when taking genistein? Researchers will compare the baseline, under treatment and washout period triglyceride, hsCRP to see if genistein works to decrease inflammation.

Participants will:

Take genistein every day for 3 months with a fixed dose manner. Afterwards, there will be 3 months washout period.

Visit the clinic once every month for checkups and tests. Keep a diary of their symptoms.

DETAILED DESCRIPTION:
Background Current medical treatment for slowing the progression of atherosclerosis focus on lipid control and anti-platelet agent use. Systemic inflammation is associated with an increased risk of cardiovascular events, independent of the cholesterol level. Recent studies showed that anti-inflammatory therapy with canakinumab or colchicine led to a significantly lower rate of recurrent cardiovascular events than placebo, independent of lipid-level lowering. Genistein was reported to be associated with anti-inflammatory and lipid lowering effects in preclinical studies. Thus, we hypothesized that genistein could provide a beneficial effect to show lipid lowering effect and anti-inflammatory effects and slow the progression of atherosclerosis.

Method The study is a phase 2 sing-center, dose-escalation clinical trial to evaluate the benefit of genistein compared to placebo among stable post-MI patients receiving standard of care therapy who have been selected for an elevated inflammatory burden as determined by high sensitivity C-reactive protein (hsCRP) > 0.1 mg/dL

Screening will take place no earlier than 28 days after the index MI and on stable (at least 4 weeks) long term medication. Evaluations will include hsCRP and determination of cancer, tuberculosis status among other measurements and procedures and will be done at a cardiology clinic. For patients who underwent percutaneous coronary intervention (PCI) at different hospital admission than the qualifying MI; screening can be initiated no earlier than 28 days following this procedure.

Intervention Patients will be screened for suitability of genistein treatment, and the trial would be initiated after informed consent. After initiation, the patients will receive genistein 250mg BID orally for complete 3 months. Afterwards, there will be 3 months washout period. Patients would then be followed for outcome measurement.

Follow-up Laboratory data would be checked 0, 1, 3, 6 months as well as clinics follow-up. Echocardiography and 6-minute walking test will be checked at 0, 3 months. Major cardiovascular event, defined as nonfatal myocardial infarction, nonfatal stroke, hospitalization for unstable angina, an arterial revascularization procedure, hospitalization for heart failure, or confirmed death from cardiovascular causes will be documented. Further follow-up would be arranged according to local guidelines until 2027/12/31 then according to patient's condition and local medical guidance.

ELIGIBILITY:
Inclusion criteria

1. Written informed consent.
2. Age ≥ 18 years.
3. History of spontaneous myocardial infarction at least 28 days before recruitment.
4. hsCRP ≥ 0.1 mg/dL
5. BMI ≥ 27

Exclusion criteria

1. Pregnant or nursing (lactating) women
2. Women of child-bearing potential
3. Planned coronary revascularization (PCI or CABG)
4. Major non-cardiac surgical or endoscopic procedure within past 6 months
5. Symptomatic patients with Class IV heart failure (HF) (New York Heart Association [NYHA].
6. Uncontrolled hypertension
7. Uncontrolled diabetes
8. History or evidence of active tuberculosis (TB) infection
9. Patients with prior history of carotid angioplasty, stenting, or carotid atherectomy
10. BMI > 40 kg/m2
11. Active cancer under treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change of triglyceride | at 3 months
  Reduction of triglyceride level from baseline at 3 months.

SECONDARY OUTCOMES:
Laboratory and functional assessment | at 1,3,6 months
  Lipid profile including total cholesterol(mg/dL), LDL-C(mg/dL), HDL-C(mg/dL), triglyceride(mg/dL) and hsCRP, HOMA-IR, TNF-alpha, IL-6
Echocardiographic assessment of ventricular function | at 1,3,6 months
  echocardiographic feature of chamber function including left ventricular ejection fraction(%), left ventricular internal diameter in end diastole (cm), left atrium dimension (mm)
Functional assessment | at 1,3,6 months
  6-minute walking test (m)

OTHER OUTCOMES:
Safety outcome | At every follow-up through study completion, with an estimated average of 1 year
  Patient reported symptoms including allergic reaction

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No